CLINICAL TRIAL: NCT04978558
Title: Cerebrovascular Autoregulation During Major Non-cardiac Surgery - a Comparison Between Near Infrared Spectroscopy and Transcranial Doppler Sonography
Brief Title: NIRS vs TCD for Cerebrovascular Autoregulation During Non-cardiac Surgery
Acronym: SONICA
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: SONICA
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cerebrovascular Circulation
Keywords: postoperative neurocognitive disorders; postoperative delirium; near-infrared spectroscopy; transcranial Doppler sonography; non-cardiac surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Continuous assessment of cerebrovascular autoregulation with NIRS and TCD — Continuous monitoring of MAP, cerebral oxygenation, and cerebral blood flow velocity before, during, and after surgery to calculate two cerebrovascular autoregulation indices Cox and Mx.

SUMMARY:
Postoperative neurocognitive disorders (NCD) are of high priority in perioperative management. The risk of suffering from NCD after surgery may be increased due to perioperative impairment of cerebrovascular autoregulation and thereby inadequate cerebral perfusion. Cerebrovascular autoregulation refers to the ability of cerebral arterioles to ensure constant cerebral blood flow independently of fluctuations in systemic blood pressure.

Cerebrovascular autoregulation can be measured based on mean arterial pressure (MAP) and a surrogate for cerebral blood flow using the correlation method. Until today, measurement of cerebral blood flow velocity assessed with transcranial Doppler sonography (TCD) is most commonly used as a non-invasive surrogate for cerebral blood flow. Alternatively, cerebral oxygenation measured with near-infrared spectroscopy (NIRS) can be used as another surrogate.

The study includes three substudies:

1. To compare NIRS and TCD for the assessment of perioperative cerebrovascular autoregulation in patients undergoing major non-cardiac surgery with an increased risk of bleeding.
2. To compare MAP for optimal cerebrovascular autoregulation before induction of general anesthesia with MAP for optimal cerebrovascular autoregulation during or after general anesthesia.
3. To analyze the association between the time-weighted average MAP below the MAP for optimal cerebrovascular autoregulation and postoperative NCD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective surgery with a minimum duration of 120 minutes
* General anesthesia
* expected blood loss > 500 ml

Exclusion Criteria:

* Temporal bone window failure (substudy 1)
* Cerebrovascular disease
* Cardiac surgery
* Neurosurgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for non-cardiac surgery with general anesthesia at a tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Equivalence of NIRS-based and TCD-based intraoperative measurement of cerebrovascular autoregulation | up to 4 hours during surgery
  calculation of cerebral autoregulation indices based on near-infrared spectroscopy and transcranial Doppler sonography
optimal MAP during NIRS-based measurement of cerebrovascular autoregulation | up to 2 hours after surgery
  MAP at lowest cerebral autoregulation index COx
delirium and postoperative NCD after surgery (composite) | days 1 to 4 after surgery (delirium), day 7 after surgery or at day of discharge from hospital (NCD)
  screening for postoperative delirium; neuropsychological testing for the assessment of cognitive function

SECONDARY OUTCOMES:
optimal MAP during TCD-based measurement of cerebrovascular autoregulation | up to 4 hours during surgery
  MAP at lowest cerebral autoregulation index (Mx)
postoperative delirium between day 1 and 4 after surgery | days 1 to 4 after surgery
  screening for postoperative delirium
delayed neurocognitive recovery at day 7 after surgery or before hospital discharge | day 7 after surgery or at day of discharge from hospital
  neuropsychological assessment
length of hospital stay | date of discharge from hospital (up to 30 days)
  duration of hospital stay (in days) between surgery and discharge
length of ICU stay | date of discharge from ICU (up to 30 days)
  duration of intensive care unit stay (in days) between surgery and discharge
mortality at 3 months after surgery | 3 months after surgery
  survival status three months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fischer, MD, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No